CLINICAL TRIAL: NCT04015024
Title: Phase IIa Clinical Study of SKLB1028 Capsule in the Treatment of FLT3 Mutation Recurrence / Refractory AML Patients
Brief Title: A Clinical Study of SKLB1028 Capsule in the Treatment of Recurrence/Refractory AML Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1028201901/PRO
Record Dates: First submitted 2019-05-22; First posted 2019-07-10 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; monotherapy; SKLB1028
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — SKLB1028; BID protein, human

STUDY DESIGN:
Intervention Model Description: The dose was initiated at 150 mg bid and after completion of the safety tolerance,200 mg bid was performed.300mg qd is safe and tolerant at phase 1 ,so the other participants were able to conduct the 300 mg qd test group when the safety tolerance.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SKLB1028 150mg bid (Experimental): Repeated oral administration until there is no longer clinical benefit from therapy,or until unacceptable toxicity occurs.
  Interventions: Drug: SKLB1028 150mg bid
- SKLB1028 200mg bid (Experimental): Repeated oral administration until there is no longer clinical benefit from therapy,or until unacceptable toxicity occurs
  Interventions: Drug: SKLB1028 200mg bid
- SKLB1028 300mg qd (Experimental): Repeated oral administration until there is no longer clinical benefit from therapy,or until unacceptable toxicity occurs
  Interventions: Drug: SKLB1028 300mg qd

INTERVENTIONS:
Drug: SKLB1028 150mg bid — 150mg oral administration twice a day
  Arms: SKLB1028 150mg bid
Drug: SKLB1028 200mg bid — 200mg oral administration twice a day
  Arms: SKLB1028 200mg bid
Drug: SKLB1028 300mg qd — 300mg oral administration once a day
  Arms: SKLB1028 300mg qd

SUMMARY:
Patients will receive oral SKLB1028 for 28 days as a course of treatment, and then to evaluate the side effects,tolerability and best dose for treating relapsed or refractory acute myeloid leukemia With FLT3 Mutations.

DETAILED DESCRIPTION:
It is an open,multicenter,queue extension study designed to characterize the efficacy and safety of different administration regimens of SKLB1028 capsules in patients with recurrent/refractory acute myeloid leukemia with FLT3 mutation. Divided into three dose groups,150mg BID,200mg BID,300mg QD. The main end point is total remission rate (ORR), total survival time (OS), progress-free survival time (PFS), remission duration, FLT3 suppression rate, competitive parameters, safety (incidence of adverse events).

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer and sign informed consent forms
2. Male or female Chinese patients, age ≥ 18 years old
3. In patients with primary or secondary aml diagnosed according to (who) classification of the World Health Organization, patients with FLT3 mutation were detected by leukemia cell gene, and refractory aml; after at least one cycle of induction treatment of: a) met any of the following conditions. B) recurrent aml; after at least one cycle of induction therapy
4. Ecog score 0-3
5. Expected survival time greater than 3 months
6. The study drug was at least 2 weeks apart from prior cytotoxic chemotherapy (except for hydroxyl groups), or at least 5 half-lives or 4 weeks with prior non-cytotoxic chemotherapy agents, short-term
7. Upper limit of normal value of serum creatinine ≤ 1.5 times
8. The upper limit of the normal value of total bilirubin ≤ 1.5 times, except for gilbert's syndrome and leukemia involving organs.
9. Upper limit of serum AST,ALT ≤ 3.0 times normal value, except where leukemia involves organs
10. The subjects of childbearing age agreed to take effective contraceptives during the treatment and 6 months after the completion of the treatment.

Exclusion Criteria:

1. Diagnosed acute promyelocytic leukemia
2. Recent symptomatic central neurosystemic leukemia
3. There are grade 2 or more non-hematological toxicity caused by previous chemotherapy
4. Bone marrow transplants within 100 days of the study
5. Uncontrollable active infections (acute or chronic fungi, bacteria, viruses, or other infections)
6. Major surgical treatment of major organs was performed in the first 4 weeks of the study
7. Radiotherapy was performed within 4 weeks before entering the study
8. Cardiac ejection fraction below 50% or below the lower limit of normal value; patients with prolonged history of qtc (male > 450 Ms, female > 470ms); severe history of heart
9. Hiv positive
10. Active hepatitis B virus infection (hepatitis B virus surface antigen positive and hepatitis B dna quantity ≥ 1 × 10^3copies/ml), hepatitis C virus infection or other liver diseases
11. Pregnant or lactating women
12. There are serious diseases or complications, or diseases that the researchers determine may endanger the safety of the patient or interfere with the study
13. Patients who are not considered to be able to enter the study
14. Treatment is currently under way in another clinical trial or in another clinical trial within four weeks of the commencement of SKLB1028 treatment
15. Patients who have previously received sklb1028 or other FLT3 inhibitors (midostaurin,gilteritinib, quizartinib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Total remission rate (ORR) | Evaluation at the end of each cycle(a cycle is 28 days) of administration and at the end of the study (assessed up to approximately 24 months)
  Complete remission (CR) + CR with incomplete hematologic recovery (CRi) + complete molecular remission (CRm) + partial remission（PR）

SECONDARY OUTCOMES:
Progression-free survival time (PFS) | Up to a total of 24 months after first dose or until disease progression, withdrawal from study, or death
Total survival time (OS) | 30 days after last subject discontinues treatment (assessed up to approximately 24 months)
CR mitigation duration (DoR-CR) | Time from the date at which the patient's objective status is first noted to be a CR to the earliest date progression is documented (assessed up to approximately 24 months
FLT3 inhibition rate | Evaluation when the patient's efficacy was evaluated as CR (assessed up to approximately 24 months)
Incidence of adverse events | From the start of the study treatment to the end of the study treatment(Within 4 weeks after the last administration)
Vital signs | From the start of the study treatment to the end of the study treatment(Within 4 weeks after the last administration)
12-lead ECG | From the start of the study treatment to the end of the study treatment(Within 4 weeks after the last administration)
physical examination | From the start of the study treatment to the end of the study treatment(Within 4 weeks after the last administration)
laboratory examination | From the start of the study treatment to the end of the study treatment(Within 4 weeks after the last administration)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China